CLINICAL TRIAL: NCT04896996
Title: The Effect of Continuous Egg Supplement on Personalized Nutri-omics in Primary School Children (SI-EGG STUDY)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 120/2560(EC2)
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Malnutrition, Child
Keywords: malnutrition; whole egg consumption; primary school student; growth
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition

STUDY DESIGN:
Intervention Model Description: A randomized controlled cluster trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whole eggs (WE) (Experimental): consume 10 additional eggs per week
  Interventions: Dietary Supplement: whole eggs
- Egg substitute (ES) (Experimental): consume the yolk-free egg substitute equivalent to 10 eggs per week
  Interventions: Dietary Supplement: yolk-free egg substitutes
- Control group (No Intervention): Regular school meals

INTERVENTIONS:
Dietary Supplement: whole eggs — whole eggs
  Arms: Whole eggs (WE)
Dietary Supplement: yolk-free egg substitutes — yolk-free egg substitutes
  Arms: Egg substitute (ES)

SUMMARY:
This research compares the effects of one-year continuous whole egg supplement vs. egg yolk substitutes and control on anthropometry, biochemical blood parameters, metabolic enzymes and microbiome data in primary school children.

DETAILED DESCRIPTION:
This research study determine the long-term effects of egg supplementation on growth, blood lipoproteins, blood proteins, nutritional status, metabolic enzymes and microbiomes in children, enrolling in the school lunch program.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 8-14 years

Exclusion Criteria:

1. Allergic of eggs
2. People who cannot continue to follow up the protocol

4. Having contra-indication i.e. problems with blood clotting

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 635 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
changes in body weight following the dietary intervention | week 0 (baseline), week 13 - 14, week 34 - 35
  weight (kg), weight for age (z-score) analysis
changes in height following the dietary intervention | week 0 (baseline), week 13 - 14, week 34 - 35
  height (cm), height for age (z-score) analysis
change in blood protein levels following dietary intervention | week 0 (baseline), week 13 - 14, week 34 - 35
  transferrin (mg/dl), pre-albumin (mg/dl), albumin (g/dl) analysis
changes in blood biochemistries following dietary intervention | week 0 (baseline), week 13 - 14, week 34 - 35
  fasting blood sugar (mg/dl), cholesterol (mg/dl), triglyceride (mg/dl), HDL-Cholesterol (mg/dl), LDL-Cholesterol (mg/dl)

SECONDARY OUTCOMES:
changes in microbioma and stool metabolites following dietary intervention | week 0 (baseline), week 13 - 14, week 34 - 35
  bacterial type, fatty acids in stool
changes in blood biochemistries following dietary intervention metabolite enzyme | week 0 (baseline), week 13 - 14, week 34 - 35
  lecithin-cholesterol acyltransferase (LCAT), cholesterol ester transfer protein (CETP), apolipoprotein C (APOC), apolipoprotein E (APOE)

CONTACTS AND LOCATIONS:
Overall Officials: Sophida Suta, MS., Study Director — Population Health and Nutrition Research Group, Siriraj Hospital, Mahidol University, Thailand
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mayurasakorn K, Sitphahul P, Hongto PO. Supplement of three eggs a week improves protein malnutrition in Thai children from rural areas. J Med Assoc Thai. 2010 Mar;93(3):301-9. PMID 20420104